CLINICAL TRIAL: NCT05852340
Title: A PHASE 1, RANDOMIZED, OPEN-LABEL, CROSSOVER STUDY TO ESTIMATE THE RELATIVE BIOAVAILABILITY OF PEDIATRIC RITLECITINIB (PF-06651600) SPRINKLED IN APPLESAUCE, YOGHURT AND STRAWBERRY JAM RELATIVE TO INTACT BLEND-IN CAPSULE OF RITLECITINIB AND THE EFFECT OF FOOD ON THE BIOAVAILABILITY OF THE INTACT BLEND-IN CAPSULE DOSAGE FORMULATION OF RITLECITINIB IN HEALTHY ADULT PARTICIPANTS
Brief Title: A Study to Assess Two Forms of The Study Medicine (Ritlecitinib) in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: B7981078; 2022-502872-22-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2023-05-01; First posted 2023-05-10 (Actual); Results first posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Healthy Volunteers; Adult; Pharmacokinetics
Keywords: Adult; Pharmacokinetic
MeSH Terms: interventions — PF-06651600

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Treatment A (Active Comparator): ritlecitinib 1 x 30 milligram (mg) intact blend-in-capsule (BiC) in fasted state
  Interventions: Drug: Ritlecitinib
- Treatment B (Active Comparator): contents of ritlecitinib 1 x 30 mg intact BiC sprinkled on strawberry jam in fasted state
  Interventions: Drug: Ritlecitinib
- Treatment C (Active Comparator): contents of ritlecitinib 1 x 30 mg intact BiC sprinkled on yoghurt in fasted state
  Interventions: Drug: Ritlecitinib
- Treatment D (Active Comparator): contents of ritlecitinib 1 x 30 mg intact BiC sprinkled on applesauce in fasted state
  Interventions: Drug: Ritlecitinib
- Treatment E (Active Comparator): ritlecitinib 1 x 30 mg intact BiC given with high fat meal
  Interventions: Drug: Ritlecitinib

INTERVENTIONS:
Drug: Ritlecitinib — ritlecitinib 1 x 30 mg intact BiC (Treatment Arms A, E)
  ritlecitinib 1 x 30 mg intact BiC sprinkled on soft foods (Treatment Arms B, C, D)
  Other Names: PF-06651600

SUMMARY:
The purpose of this study is to compare if two forms of study medicine, Ritlecitinib, get processed differently in healthy adults.

This study is seeking participants who are:

* aged 18 or older;
* male or female who are healthy as determined by medical assessment ;
* Body-mass Index (BMI) of 16 to 32, and a total body weight > 45kg.

The study will take up to 2.5 months, including the screening period. There will be 5 periods in total for this study. Participants will have to stay at the study clinic for at least 11 days. Participants will take Riltecitinib either as sprinkled in Soft Food or as Intact Blend-In Capsule. On day 1 of each period, participants will take Riltecitinib and have blood samples taken both before and afterwards. Participants will also answer questions for taste assessment purpose. A follow-up phone call will be made at 28 to 35 days after the last study period.

DETAILED DESCRIPTION:
Ritlecitinib is a covalent and irreversible inhibitor of JAK3 with high selectivity over the other JAK isoforms (JAK1, JAK2, and TYK2). Ritlecitinib also inhibits irreversibly the tyrosine kinase expressed in TEC family kinases with selectivity over the broader human kinome. Treatment with ritlecitinib is expected to inhibit the inflammatory pathways mediated by IL 7, IL 15 and IL 21, all implicated in UC, CD, AA, RA, and vitiligo. Moreover, due to lack of activity against the other JAK isoforms, ritlecitinib is expected to spare immunoregulatory cytokines such as IL 10, IL 27 and IL 35, which are critical to the maintenance of immunosuppressive functions and immune homeostasis.

The objective of this study is to estimate the impact of administration methods on the bioavailability of the pediatric ritlecitinib intact BiC formulation. The study will be conducted as a Phase 1, open-label, single dose, randomized, 4-crossover periods and 1-fixed period design in a single cohort of approximately 12 healthy male or female participants at a single center. Participants will be randomized into 1 of 4 sequences of treatment. Blood samples will be collected for PK analysis. A taste assessment will be also conducted.

Participants will participate in the study for up to approximately 2.5 months, with the inclusion of the screening and follow-up period. On Day 1 of each period, participants will receive a single dose of IP. Administration of IP will be via dosing using intact BiCs with water or by emptying the capsule contents on soft food as per dosing instructions.

Participants will be confined in the CRU for a total of at least 11 days and discharged at the discretion of the investigator. A follow-up phone call will be made at least 28 calendar days and up to 35 calendar days after the last administration of the study intervention to capture any potential AE and confirm appropriate contraceptive usage.

Tolerability and safety will be assessed for all treatments by monitoring AEs.

ELIGIBILITY:
Key Inclusion Criteria:

1. Aged 18 or older.
2. Male or female who are healthy as determined by medical assessment.
3. Body-mass Index (BMI) of 16 to 32, and a total body weight > 45kg.

Key Exclusion Criteria:

1. Any condition possibly affecting drug absorption (eg, gastrectomy, cholecystectomy).
2. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
3. Known immunodeficiency disorder, including positive serology for HIV, or a first degree relative with a hereditary immunodeficiency, or infections (acute or chronic).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-05-09 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-07-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit - Brussels, Brussels, Bruxelles-capitale, Région de, Belgium

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7981078

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This is a phase 1, open-label, single dose, randomized 4-crossover periods (periods 1-4) and 1-fixed period (period 5) design study. A total of 12 participants were randomized and assigned to receive the study intervention.
Groups:
- Sequence 1: Treatment A-> B-> C-> D-> E: Participants were randomized to receive ritlecitinib 30 milligram (mg) intact blend-in capsule (BiC) in fasted state on Day 1 of Period 1 (Treatment A). Period 1 was followed by Period 2. On Day 1 of Period 2, participants received contents of ritlecitinib 30 mg BiC sprinkled on strawberry jam in fasted state (Treatment B). Period 2 was followed by Period 3. On Day 1 of Period 3, participants received contents of ritlecitinib 30 mg BiC sprinkled on yoghurt in fasted state (Treatment C). Period 3 was followed by Period 4. On Day 1 of Period 4, participants received contents of ritlecitinib 30 mg BiC sprinkled on applesauce in fasted state (Treatment D). Period 4 was followed by Period 5. On Day 1 of Period 5, participants received ritlecitinib 30 mg intact BiC given with high fat meal (Treatment E). Dosing of each period was separated by at least a 48-hour washout interval. Participants were followed up for up to 35 days after the last administration of ritlecitinib.
- Sequence 2: Treatment B-> D-> A-> C-> E: Participants were randomized to receive contents of ritlecitinib 30 mg BiC sprinkled on strawberry jam in fasted state on Day 1 of Period 1 (Treatment B). Period 1 was followed by Period 2. On Day 1 of Period 2, participants received contents of ritlecitinib 30 mg BiC sprinkled on applesauce in fasted state (Treatment D). Period 2 was followed by Period 3. On Day 1 of Period 3, participants received ritlecitinib 30 mg intact BiC in fasted state (Treatment A). Period 3 was followed by Period 4. On Day 1 of Period 4, participants received contents of ritlecitinib 30 mg BiC sprinkled on yoghurt in fasted state (Treatment C). Period 4 was followed by Period 5. On Day 1 of Period 5, participants received ritlecitinib 30 mg intact BiC given with high fat meal (Treatment E). Dosing of each period was separated by at least a 48-hour washout interval. Participants were followed up for up to 35 days after the last administration of ritlecitinib.
- Sequence 3: Treatment C-> A-> D-> B-> E: Participants were randomized to receive contents of ritlecitinib 30 mg BiC sprinkled on yoghurt in fasted state on Day 1 of Period 1 (Treatment C). Period 1 was followed by Period 2. On Day 1 of Period 2, participants received ritlecitinib 30 mg intact BiC in fasted state (Treatment A). Period 2 was followed by Period 3. On Day 1 of Period 3, participants received contents of ritlecitinib 30 mg BiC sprinkled on applesauce in fasted state (Treatment D). Period 3 was followed by Period 4. On Day 1 of Period 4, participants received contents of ritlecitinib 30 mg BiC sprinkled on strawberry jam in fasted state (Treatment B). Period 4 was followed by Period 5. On Day 1 of Period 5, participants received ritlecitinib 30 mg intact BiC given with high fat meal (Treatment E). Dosing of each period was separated by at least a 48-hour washout interval. Participants were followed up for up to 35 days after the last administration of ritlecitinib.
- Sequence 4: Treatment D-> C-> B-> A-> E: Participants were randomized to receive contents of ritlecitinib 30 mg BiC sprinkled on applesauce in fasted state on Day 1 of Period 1 (Treatment D). Period 1 was followed by Period 2. On Day 1 of Period 2, participants received contents of ritlecitinib 30 mg BiC sprinkled on yoghurt in fasted state (Treatment C). Period 2 was followed by Period 3. On Day 1 of Period 3, participants received contents of ritlecitinib 30 mg BiC sprinkled on strawberry jam in fasted state (Treatment B). Period 3 was followed by Period 4. On Day 1 of Period 4, participants received ritlecitinib 30 mg intact BiC in fasted state (Treatment A). Period 4 was followed by Period 5. On Day 1 of Period 5, participants received ritlecitinib 30 mg intact BiC given with high fat meal (Treatment E). Dosing of each period was separated by at least a 48-hour washout interval. Participants were followed up for up to 35 days after the last administration of ritlecitinib.
Period: Period 1
Arm/Group | Sequence 1: Treatment A-> B-> C-> D-> E | Sequence 2: Treatment B-> D-> A-> C-> E | Sequence 3: Treatment C-> A-> D-> B-> E | Sequence 4: Treatment D-> C-> B-> A-> E
Started | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | Sequence 1: Treatment A-> B-> C-> D-> E | Sequence 2: Treatment B-> D-> A-> C-> E | Sequence 3: Treatment C-> A-> D-> B-> E | Sequence 4: Treatment D-> C-> B-> A-> E
Started | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | Sequence 1: Treatment A-> B-> C-> D-> E | Sequence 2: Treatment B-> D-> A-> C-> E | Sequence 3: Treatment C-> A-> D-> B-> E | Sequence 4: Treatment D-> C-> B-> A-> E
Started | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0
Period: Period 4
Arm/Group | Sequence 1: Treatment A-> B-> C-> D-> E | Sequence 2: Treatment B-> D-> A-> C-> E | Sequence 3: Treatment C-> A-> D-> B-> E | Sequence 4: Treatment D-> C-> B-> A-> E
Started | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0
Period: Period 5
Arm/Group | Sequence 1: Treatment A-> B-> C-> D-> E | Sequence 2: Treatment B-> D-> A-> C-> E | Sequence 3: Treatment C-> A-> D-> B-> E | Sequence 4: Treatment D-> C-> B-> A-> E
Started | 3 | 3 | 3 | 3
Completed | 3 | 2 | 3 | 2
Not Completed | 0 | 1 | 0 | 1
Not completed — Not completing the meal | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants who were enrolled in the study.
Groups:
- All Participants: All participants who were enrolled in the study.
Arm/Group | All Participants
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.4 (12.99)
Age, Customized [Count of Participants; unit: Participants]
  26-35 years | 6
  36-45 years | 3
  >45 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-Time Profile From Time Zero Extrapolated to Infinite Time (AUCinf) of Ritlecitinib
Description: AUCinf was defined as area under the plasma-concentration time profile from time zero extrapolated to infinite time. AUCinf for ritlecitinib was calculated by AUClast + (Clast/kel), where Clast was the predicted plasma concentration at the last quantifiable time point from the log-linear regression analysis and kel was the terminal phase rate constant calculated by a linear regression of the log-linear concentration time curve.
Time Frame: 0 (pre-dose), 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12 and 24 hours post-dose on Day 1 of each period. Each treatment period lasted 24 hours. Dosing of each period was separated by at least a 48-hour washout interval.
Population: All participants randomized and treated who had at least 1 of the pharmacokinetic (PK) parameters of primary interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Groups:
- Ritlecitinib 30 mg Capsule (Fasted): Participants received a single oral dose of ritlecitinib 30 mg capsule under fasted conditions on Day 1 of each Period.
- Ritlecitinib 30 mg Capsule Mixed With Strawberry Jam (Fasted): Participants received a single oral dose of ritlecitinib 30 mg capsule mixed with strawberry jam under fasted conditions on Day 1 of each Period.
- Ritlecitinib 30 mg Capsule Mixed With Yoghurt (Fasted): Participants received a single oral dose of ritlecitinib 30 mg capsule mixed with yoghurt under fasted conditions on Day 1 of each Period.
- Ritlecitinib 30 mg Capsule Mixed With Applesauce (Fasted): Participants received a single oral dose of ritlecitinib 30 mg capsule mixed with applesauce under fasted conditions on Day 1 of each Period.
- Ritlecitinib 30 mg Capsule Given With High Fat Meal: Participants received a single oral dose of ritlecitinib 30 mg capsule given with high fat meal on Day 1 of each Period.
Arm/Group | Ritlecitinib 30 mg Capsule (Fasted) | Ritlecitinib 30 mg Capsule Mixed With Strawberry Jam (Fasted) | Ritlecitinib 30 mg Capsule Mixed With Yoghurt (Fasted) | Ritlecitinib 30 mg Capsule Mixed With Applesauce (Fasted) | Ritlecitinib 30 mg Capsule Given With High Fat Meal
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 9
nanogram*hour per milliliter (ng*hr/mL) | 389.1 (32) | 398.3 (31) | 378.0 (27) | 387.8 (27) | 387.0 (23)
Statistical Analysis 1: Comparison: Ritlecitinib 30 mg Capsule (Fasted) vs Ritlecitinib 30 mg Capsule Mixed With Strawberry Jam (Fasted); Reference: Ritlecitinib 30 mg Capsule (Fasted) Test: Ritlecitinib 30 mg Capsule Mixed with Strawberry Jam (Fasted); Test type: Other — Analysis done using a mixed effect model with sequence, period and treatment as fixed effects and participant within sequence as a random effect. Ratio (Test/Reference) and 90% confidence interval (CI) are expressed as percentages; Ratio (%) of Adjusted Geometric Means = 102.36, 90% CI 2-sided [95.81 to 109.35]
Statistical Analysis 2: Comparison: Ritlecitinib 30 mg Capsule (Fasted) vs Ritlecitinib 30 mg Capsule Mixed With Yoghurt (Fasted); Reference: Ritlecitinib 30 mg Capsule (Fasted) Test: Ritlecitinib 30 mg Capsule Mixed with Yoghurt (Fasted); Test type: Other — Analysis done using a mixed effect model with sequence, period and treatment as fixed effects and participant within sequence as a random effect. Ratio (Test/Reference) and 90% CI are expressed as percentages; Ratio (%) of Adjusted Geometric Means = 97.15, 90% CI 2-sided [90.94 to 103.79]
Statistical Analysis 3: Comparison: Ritlecitinib 30 mg Capsule (Fasted) vs Ritlecitinib 30 mg Capsule Mixed With Applesauce (Fasted); Reference: Ritlecitinib 30 mg Capsule (Fasted) Test: Ritlecitinib 30 mg Capsule Mixed with Applesauce (Fasted); Test type: Other — [test comment as in outcome 1, analysis 2]; Ratio (%) of Adjusted Geometric Means = 99.65, 90% CI 2-sided [93.28 to 106.46]
Statistical Analysis 4: Comparison: Ritlecitinib 30 mg Capsule (Fasted) vs Ritlecitinib 30 mg Capsule Given With High Fat Meal; Reference: Ritlecitinib 30 mg Capsule (Fasted) Test: Ritlecitinib 30 mg Capsule Given with High Fat Meal; Test type: Other — [test comment as in outcome 1, analysis 2]; Ratio (%) of Adjusted Geometric Means = 104.84, 90% CI 2-sided [97.30 to 112.96]

2. Primary Outcome: Maximum Observed Concentration (Cmax) of Ritlecitinib
Description: Cmax was defined as maximum observed plasma concentration. Cmax for ritlecitinib was observed directly from data.
Time Frame: as for outcome 1
Population: All participants randomized and treated who had at least 1 of the PK parameters of primary interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Ritlecitinib 30 mg Capsule (Fasted) | Ritlecitinib 30 mg Capsule Mixed With Strawberry Jam (Fasted) | Ritlecitinib 30 mg Capsule Mixed With Yoghurt (Fasted) | Ritlecitinib 30 mg Capsule Mixed With Applesauce (Fasted) | Ritlecitinib 30 mg Capsule Given With High Fat Meal
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 10
ng/mL | 244.3 (35) | 236.1 (28) | 206.6 (24) | 229.4 (25) | 108.0 (28)
Statistical Analysis 1: Comparison: Ritlecitinib 30 mg Capsule (Fasted) vs Ritlecitinib 30 mg Capsule Mixed With Strawberry Jam (Fasted); Reference: Ritlecitinib 30 mg Capsule (Fasted) Test: Ritlecitinib 30 mg Capsule Mixed with Strawberry Jam (Fasted); Test type: Other — [test comment as in outcome 1, analysis 2]; Ratio (%) of Adjusted Geometric Means = 96.63, 90% CI 2-sided [83.66 to 111.62]
Statistical Analysis 2: Comparison: Ritlecitinib 30 mg Capsule (Fasted) vs Ritlecitinib 30 mg Capsule Mixed With Yoghurt (Fasted); Reference: Ritlecitinib 30 mg Capsule (Fasted) Test: Ritlecitinib 30 mg Capsule Mixed with Yoghurt (Fasted); Test type: Other — [test comment as in outcome 1, analysis 2]; Ratio (%) of Adjusted Geometric Means = 84.58, 90% CI 2-sided [73.23 to 97.70]
Statistical Analysis 3: Comparison: Ritlecitinib 30 mg Capsule (Fasted) vs Ritlecitinib 30 mg Capsule Mixed With Applesauce (Fasted); Reference: Ritlecitinib 30 mg Capsule (Fasted) Test: Ritlecitinib 30 mg Capsule Mixed with Applesauce (Fasted); Test type: Other — [test comment as in outcome 1, analysis 2]; Ratio (%) of Adjusted Geometric Means = 93.91, 90% CI 2-sided [81.30 to 108.48]
Statistical Analysis 4: Comparison: Ritlecitinib 30 mg Capsule (Fasted) vs Ritlecitinib 30 mg Capsule Given With High Fat Meal; Reference: Ritlecitinib 30 mg Capsule (Fasted) Test: Ritlecitinib 30 mg Capsule Given with High Fat Meal; Test type: Other — [test comment as in outcome 1, analysis 2]; Ratio (%) of Adjusted Geometric Means = 43.83, 90% CI 2-sided [37.50 to 51.23]

3. Secondary Outcome: Number of Participants With All-Causality and Treatment-Related Treatment Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study treatment without regard to possibility of causal relationship. Treatment-related AE was any untoward medical occurrence attributed to study treatment in a participant who received study treatment. Relatedness to study treatment was assessed by the investigator. A serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent events were events between first dose of study treatment and up to approximately 35 days that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: From the first dose of study treatment up to 28-35 days after last dose of study treatment (ie, up to 45 days)
Population: All participants who took at least 1 dose of study intervention. Participants were analyzed according to the study intervention they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Ritlecitinib 30 mg Capsule (Fasted) | Ritlecitinib 30 mg Capsule Mixed With Strawberry Jam (Fasted) | Ritlecitinib 30 mg Capsule Mixed With Yoghurt (Fasted) | Ritlecitinib 30 mg Capsule Mixed With Applesauce (Fasted) | Ritlecitinib 30 mg Capsule Given With High Fat Meal
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 10
Participants
  Number of participants with all-causality TEAEs | 5 | 2 | 4 | 4 | 2
  Number of participants with all-causality SAEs | 0 | 0 | 0 | 0 | 0
  Number of participants with treatment-related TEAEs | 2 | 0 | 1 | 0 | 1
  Number of participants with treatment-related SAEs | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Number of Participants With Laboratory Abnormalities
Description: Hematology included hemoglobin, hematocrit, red blood cell count, mean corpuscular volume, mean corpuscular hemoglobin, mean corpuscular hemoglobin concentration, platelet and white blood cell count, total neutrophils, eosinophils, etc. Chemistry included blood urea nitrogen, creatinine, glucose, calcium, sodium, potassium, chloride, bicarbonate, aspartate aminotransferase, alanine aminotransferase, total bilirubin, alkaline phosphatase, uric acid, albumin, total protein, etc. Urinalysis included pH, glucose, protein, blood, ketones, nitrites, leukocyte esterase, urobilinogen, urine bilirubin and microscopy. Laboratory abnormalities were judged by the investigator. Laboratory abnormalities reported for at least 1 participant in the whole study are presented here.
Time Frame: From the first dose of study treatment up to 28-35 days after last dose of study treatment (ie, up to 45 days)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Ritlecitinib 30 mg Capsule (Fasted) | Ritlecitinib 30 mg Capsule Mixed With Strawberry Jam (Fasted) | Ritlecitinib 30 mg Capsule Mixed With Yoghurt (Fasted) | Ritlecitinib 30 mg Capsule Mixed With Applesauce (Fasted) | Ritlecitinib 30 mg Capsule Given With High Fat Meal
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 10
Participants | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From the first dose of study treatment up to 28-35 days after last dose of study treatment (ie, up to 45 days)
Arm/Group | Ritlecitinib 30 mg Capsule (Fasted) | Ritlecitinib 30 mg Capsule Mixed With Strawberry Jam (Fasted) | Ritlecitinib 30 mg Capsule Mixed With Yoghurt (Fasted) | Ritlecitinib 30 mg Capsule Mixed With Applesauce (Fasted) | Ritlecitinib 30 mg Capsule Given With High Fat Meal
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12 | 0/10
Other Adverse Events (participants affected / at risk) | 5/12 | 2/12 | 4/12 | 4/12 | 2/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ritlecitinib 30 mg Capsule (Fasted) (N=12) | Ritlecitinib 30 mg Capsule Mixed With Strawberry Jam (Fasted) (N=12) | Ritlecitinib 30 mg Capsule Mixed With Yoghurt (Fasted) (N=12) | Ritlecitinib 30 mg Capsule Mixed With Applesauce (Fasted) (N=12) | Ritlecitinib 30 mg Capsule Given With High Fat Meal (N=10)
Dry eye (Eye disorders) | 0 | 0 | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Lip dry (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 1 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2
Haematoma (Vascular disorders) | 1 | 1 | 2 | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2023-02-02): https://cdn.clinicaltrials.gov/large-docs/40/NCT05852340/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-27): https://cdn.clinicaltrials.gov/large-docs/40/NCT05852340/SAP_001.pdf